CLINICAL TRIAL: NCT05172349
Title: Pilote Study of the Use of a Double Amniotic Membrane Inserted in a Ring of Umbilical Vessels With Wharton's Jelly, Tissues Treated by the AMTRIX Process, in the Treatment of Trophic Ulcers
Brief Title: Use of a Biological Lens of Amniotic Membrane (LV-Visio-AMTRIX) in the Treatment of Trophic Ulcers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in sponsor's strategy
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-Visio-AMTRIX-TBF4; IDRCB (Registry Identifier: 2020-A00656-33)
Record Dates: First submitted 2021-12-07; First posted 2021-12-29 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Corneal Ulcer; Persistent Corneal Epithelial Defect
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LV-Visio-AMTRIX (Experimental): Sutureless amniotic membrane supported by a biological ring positioned by the investigator during patients' hospital visits.
  Interventions: Biological: LV-Visio-AMTRIX

INTERVENTIONS:
Biological: LV-Visio-AMTRIX — Chemically-treated, viro-inactivated, freeze-dried and irradiated allograft placed by the investigator during patients' hospital visit

SUMMARY:
The purpose of this open, multicenter pilot trial is to assess the impact of the use of an amniotic membrane on the healing of a persistent epithelial lesion or of a corneal ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 80 years old
* Stage 2 (persistent epithelial lesion : LEP) or stage 3 (corneal ulcer) trophic ulcer affecting only one eye. Patient whose contralateral eye is affected by stage 1 neurotrophic keratitis may also be included
* Two or more weeks old LEP or corneal ulcer refractory to one or more conventional nonsurgical therapies
* Absence of objective evidence of improvement of the epithelial ulceration or corneal ulcer within 2 weeks prior to study inclusion
* Failure of amniotic membrane treatment of the trophic ulcer: failure by absence of healing a few day after overlay treatment or 15 days after inlay grafting
* Patient able to understand French language
* Informed and consenting patient
* Patient affiliated to a social security system or beneficiary of such a system

Exclusion Criteria:

* Pregnant or breastfeeding patient or without contraception for non-menopausal women
* Active infectious ulcer
* Preperforating ulcer or ulcer that has reached the posterior 1/3 of the storm
* Allergy to Oxybuprocaine or Tetracaine eye drops, to ester type local anesthetics and to fluorescein
* Current contact lens wear, including scleral lenses
* NSAID eye drops and any drops containing preservatives
* Antibiotic, anti-viral, anti-parasitic eye drops
* Patients with identified causes of the ulcer for which medical treatment without preservatives or other healing treatment is beneficial
* Ocular surgery for other pathology than the trophic ulcer in the 3 months preceding the inclusion in the study
* Ophthalmologic pathology requiring daily eye drops
* Monophtalmic patients
* Persons deprived of liberty by a judicial or administrative decision
* Adults who are subject to a legal protection measure or who are unable to express their consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Largest diameter of persistent epithelial lesion area or corneal ulcer under 0.5 mm | 15 days
  Diameter assessed by centralized reading on photograph after fluorescein test

SECONDARY OUTCOMES:
Recovery of the visual acuity evaluated by Monoyer chart | 30 days, 45 days
Stable or decreased score for inflammatory and clinical signs of the ocular surface | 2 days, 4 days, 7 days, 10 days, 15 days, 30 days, 45 days
  Composite score for inflammatory and clinical signs of the ocular surface on 66 points. Duration and intensity are evaluated for secretion, dry eyes, tearing, foreign body sensation, fluctuating vision, photophobia, burning sensation and lids edema. Duration is evaluated from a scale from 0: never to 4: all the time. Intensity is evaluated from a scale from 0: slight to 2: severe. Localization and intensity are evaluated for conjunctival edema, conjunctival redness and neovascularization. Localization is evaluated on a scale from 0: no reaction to 4: reaction present in the whole eye.
Stabilisation or decrease of pain evaluated on visual analog scale | 2 days, 4 days, 7 days, 10 days, 15 days, 30 days, 45 days
  VAS on 10 points from 0: no pain to 10: worst imaginable pain